CLINICAL TRIAL: NCT05077930
Title: Validation Protocol for The Clinical Use of Convalescent Plasma for Hospitalized Patients With COVID-19. A Prospective Study at a Hospital in Southern Brazil.
Brief Title: Convalescent Plasma Therapy for Hospitalized Patients With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tânia Portella Costa (Other)
Collaborators: Centro de Hematologia e Hemoterapia do Paraná - Hemepar (Unknown); Fundação Oswaldo Cruz, Instituto Carlos Chagas, ICC Paraná (Unknown); Science Valley Research Institute (Other)
Responsible Party: Sponsor-Investigator, Tânia Portella Costa, Tânia Portella Costa - Maternidade e Cirurgia Nossa Senhora do Rocio/ SA - Hospital do Rocio, Science Valley Research Institute
Organization: Science Valley Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCP TRIAL
Record Dates: First submitted 2021-10-08; First posted 2021-10-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: COVID-19; Convalescent Plasma; SARS-CoV-2; Pneumonia; Coronavirus Infections; Respiratory Tract Diseases
MeSH Terms: conditions — COVID-19; Pneumonia; Coronavirus Infections; Respiratory Tract Diseases | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is an open-label, randomized study design (1: 1), controlled trial, in hospitalized patients with COVID-19.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma (Experimental): The investigational product is anti-SARS-CoV-2 convalescent plasma obtained from former patients identified as having recovered from COVID-19 and obtained by Centro de Hematologia e Hemoterapia do Paraná - Hemepar following national blood donation guidelines and Brazilian Health Regulatory Agency (ANVISA) criteria. Potential donors will be screened using an anti-SARS-CoV-2 serologic assay and antibody levels will be determined. Participants will receive the standard of care treatment and a single unit of convalescent plasma (volume=200 mL or 400 mL).
  Interventions: Biological: Convalescent plasma
- Standard of care (Active Comparator): Standard of care treatment according to the institutional protocol.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Biological: Convalescent plasma — The intervention group will receive 200 or 400 mL of high-titer COVID-19 convalescent plasma, ABO compatible with the patient, within 24 hours of randomization.
  Arms: Convalescent Plasma
Drug: Standard of care — The active comparator group will receive oxygen supplementation, corticoids, antiretrovirals, and/or monoclonal antibodies according to the institutional protocol.
  Arms: Standard of care

SUMMARY:
Plasma from donors who have recovered from coronavirus disease 2019 (COVID-19) contain antibodies to SARS-CoV-2 and may be a potential therapy for hospitalized patients with COVID-19. The efficacy of high-titer convalescent plasma for COVID-19, however, still unclear. The present study aims to evaluate the efficacy and safety of using convalescent plasma for treating hospitalized patients with COVID-19.

DETAILED DESCRIPTION:
This is an open-label, randomized controlled trial aimed to evaluate the efficacy and safety of using convalescent plasma for treating hospitalized patients with COVID-19. Participants must be adult hospitalized patients with a confirmed diagnosis of COVID-19 and time Between symptom onset and inclusion ≤ 7 days. Two hundred participants will be randomized in a 1:1 ratio to receive either 200-400 mL of high-titer COVID-19 convalescent plasma or standard care. The primary endpoint is the proportion of patients with clinical improvement at day 14 following randomization, defined by an increase of two points in the 7-point ordinal scale based on that recommended by the World Health Organization. Safety will be daily assessed by monitoring the occurrence of adverse effects and reactions to convalescent plasma transfusion. Study visits will occur on Day 1, Day 3, Day 7, and Day 14 or until hospital discharge, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients aged ≥18 years.
* Confirmed diagnosis of COVID-19 by RT-PCR or antigen test in respiratory samples.
* Time between symptom onset and inclusion ≤ 7 days.
* Enrolled within 5 days of hospitalization.
* Sign the consent form.

Exclusion Criteria:

* Contraindication to transfusion due to inability to tolerate additional fluid, such as due to decompensated congestive heart failure.
* History of previous severe allergic reactions to transfused blood products.
* Limiting comorbidity for administering the therapies provided for in this protocol in the opinion of the investigator.
* Not currently enrolled another interventional clinical trial of COVID-19 treatment.
* Critically ill patient with COVID-19 being treated in intensive care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-07 (Actual)

PRIMARY OUTCOMES:
Clinical status on a 7-point ordinal scale | From randomization to end of study at Day 14
  Patients' clinical status over time assessed by a 7-point ordinal scale from World Health Organization (WHO). Lower scores are seen with better clinical outcomes. The scale categories are as follows: (1), not hospitalized with resumption of normal activities; (2), not hospitalized, but unable to resume normal activities; (3), hospitalized, not requiring supplemental oxygen; (4), hospitalized, requiring supplemental oxygen; (5), hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation; (6), hospitalized, requiring ECMO (extracorporeal membrane oxygenation), IMV (intermittent mandatory ventilation), or both; (7), death.
  Proportion of patients with clinical improvement, defined by an increase of two points in the ordinal scale of seven WHO categories.

SECONDARY OUTCOMES:
Percentage of participants at each clinical status on a 7-point ordinal scale | Day 1, Day 3, Day 7, and Day 14 after randomization
  Measure of patients' clinical status using an ordinal scale for clinical improvement created by World Health Organization (WHO) and based on 7-point scale categories. Lower scores in this scale are seen with better clinical outcomes. The scale categories are as follows: (1), not hospitalized with resumption of normal activities; (2), not hospitalized, but unable to resume normal activities; (3), hospitalized, not requiring supplemental oxygen; (4), hospitalized, requiring supplemental oxygen; (5), hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation; (6), hospitalized, requiring ECMO, IMV, or both; (7), death.
Oxygen saturation | Day 1, Day 3, Day 7, and Day 14 after randomization
Prevalence of oxygen-intake methods | Day 1, Day 3, Day 7, and Day 14 after randomization
  Percentage of participants using oxygen by mask or nasal prongs, oxygen by non-invasive ventilation or high flow, intubation & mechanical ventilation and ECMO.
Respiratory rate | Day 1, Day 3, Day 7, and Day 14 after randomization
The PaO2 / FiO2 ratio (for patients on mechanical mechanisms) | Day 1, Day 3, Day 7, and Day 14 after randomization
Number and /or extension of affected lung areas on chest computed tomography | Day 1, Day 3, Day 7, and Day 14 after randomization
Length of hospital stay | Day 1, Day 3, Day 7, and Day 14 after randomization
Length of stay in intensive care | Day 1, Day 3, Day 7, and Day 14 after randomization
Time until independence from oxygen therapy in days | Day 1, Day 3, Day 7, and Day 14 after randomization
Ventilator free days | Day 1, Day 3, Day 7, and Day 14 after randomization
In patients who needed mechanical ventilation, time to initiate mechanical ventilation (calculated in days, from entry into the protocol until orotracheal intubation) | Day 1, Day 3, Day 7, and Day 14 after randomization
Rate of transfusion reactions to convalescent plasma infusion | Daily, until Day 14 after randomization
Percentage of participants who develop serious adverse events and adverse events considered as definitely or probably associated with plasma transfusion | Daily, until Day 14 after randomization
  Adverse events (worsening anemia, urticaria, skin rash, transfusion-associated circulatory overload, and others) assessed during hospitalization.

OTHER OUTCOMES:
Association between the presence of comorbidities at baseline and clinical status on a 7-point ordinal scale | Day 1 and Day 14 after randomization
  Association between patients' clinical status assessed by a 7-point ordinal scale from World Health Organization (WHO) on Day 14 after randomization and baseline characteristics and history or comorbidities known at high risk for COVID-19 (age, sex, obesity - body mass index >30 kg/m², history of hypertension, chronic heart disease, congestive heart failure, chronic bronchopulmonary disease, diabetes mellitus, and immunosuppression).
  Lower scores in this scale are seen with better clinical outcomes. The scale categories are as follows: (1), not hospitalized with resumption of normal activities; (2), not hospitalized, but unable to resume normal activities; (3), hospitalized, not requiring supplemental oxygen; (4), hospitalized, requiring supplemental oxygen; (5), hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation; (6), hospitalized, requiring ECMO, IMV, or both; (7), death.
Association between the volume of convalescent plasma transfused and clinical status on a 7-point ordinal scale | Day 1 and Day 14 after randomization
  Association between patients' clinical status assessed by a 7-point ordinal scale from World Health Organization (WHO) on Day 14 after randomization and the volume of a single unit of convalescent plasma transfused (200 mL or 400 mL). Lower scores in this scale are seen with better clinical outcomes. The scale categories are as follows: (1), not hospitalized with resumption of normal activities; (2), not hospitalized, but unable to resume normal activities; (3), hospitalized, not requiring supplemental oxygen; (4), hospitalized, requiring supplemental oxygen; (5), hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation; (6), hospitalized, requiring ECMO, IMV, or both; (7), death.
Changes from baseline in inflammatory surrogate markers: white blood counts, lymphocyte counts, C-reactive protein (CRP) and D-dimer levels | Day 1 and Day 14 after randomization
Association between the concentration of inflammatory surrogate markers and clinical status on a 7-point ordinal scale | Day 14 after randomization
  Association between patients' clinical status assessed by a 7-point ordinal scale from World Health Organization (WHO) on Day 14 after randomization and inflammatory surrogate markers, which include white blood counts, lymphocyte counts, C-reactive protein (CRP) and D-dimer levels. Lower scores in this scale are seen with better clinical outcomes. The scale categories are as follows: (1), not hospitalized with resumption of normal activities; (2), not hospitalized, but unable to resume normal activities; (3), hospitalized, not requiring supplemental oxygen; (4), hospitalized, requiring supplemental oxygen; (5), hospitalized, requiring high-flow oxygen therapy or noninvasive mechanical ventilation; (6), hospitalized, requiring ECMO, IMV, or both; (7), death.

CONTACTS AND LOCATIONS:
Overall Officials: Kengi Itinose, MD, Study Director — Maternidade e Cirurgia Nossa Senhora do Rocio/ SA - Hospital do Rocio
Locations (1):
- Maternidade e Cirurgia Nossa Senhora do Rocio/ SA - Hospital do Rocio, Campo Largo, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piechotta V, Chai KL, Valk SJ, Doree C, Monsef I, Wood EM, Lamikanra A, Kimber C, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Jul 10;7(7):CD013600. doi: 10.1002/14651858.CD013600.pub2. PMID 32648959
- [Derived] Costa TP, Aoki M, Ribeiro CM, Socca E, Itinose L, Basso R, Blanes L. Efficacy of convalescent plasma in hospitalized COVID-19 patients: findings from a controlled trial. Braz J Med Biol Res. 2024 Oct 7;57:e13627. doi: 10.1590/1414-431X2024e13627. eCollection 2024. PMID 39383382
- See also: Core Outcome Set (COS) for studies of any intervention in hospitalised patients with confirmed or suspected COVID-19 — https://www.comet-initiative.org/assets/downloads/COVID-19%20meta%20COS_Table%201_15th%20March%202021.pdf